CLINICAL TRIAL: NCT01712867
Title: The Effect of Phytosterol Esters of Omega-3 (Vayarol) Versus Omega-3 Acids Ethyl Esters in Reducing Triglyceride Levels in Hypertriglyceridemia Patients: A Double-blind, Randomized, Noninferiority Trial
Brief Title: The Effect of Phytosterol Esters of Omega-3 (Vayarol) Versus Omega-3 Acids Ethyl Esters in Reducing Triglyceride Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Enzymotec (Industry)
Collaborators: Daewon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Vayarol_006
Record Dates: First submitted 2012-10-18; First posted 2012-10-24 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Patients With Hypertriglyceridemia
MeSH Terms: interventions — Omacor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Phytosterol esters of omega-3 (Experimental): 4 capsules/day for 12 weeks
  Interventions: Other: Phytosterol esters of omega-3
- Omega-3 acid ethyl esters (Active Comparator): 4 capsules/day for 12 weeks
  Interventions: Other: Omega-3 acid ethyl esters

INTERVENTIONS:
Other: Omega-3 acid ethyl esters — 4 capsules/day for 12 weeks
  Arms: Omega-3 acid ethyl esters
Other: Phytosterol esters of omega-3 — 4 capsules/day for 12 weeks
  Arms: Phytosterol esters of omega-3

SUMMARY:
The primary objective is to determine the efficacy of phytosterol esters of omega-3 (Vayarol) versus Omega-3 acids ethyl esters in reducing triglyceride levels in hypertriglyceridemia patients with fasting triglyceride levels ≥ 200 and < 500 mg/dL.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age > 18 years
2. Triglycerides ≥ 200 mg/dL and < 500 mg/dL
3. Ability to give written informed consent

Exclusion Criteria:

1. Female patient who are pregnant or breastfeeding or planning to become pregnant
2. Fasting plasma glucose (FPG) levels > 110 mg/dL
3. Type 2 diabetes mellitus that is poorly controlled (glycosylated hemoglobin [HbAlc ] >8.0%
4. Patients who are under use of lipid altering drugs excluding use of Simvastatin, Atorvastatin, and Rosovastatin for 6 weeks or more
5. Patients who are under use of products containing omega-3 fatty acids or other dietary supplements with potential lipid altering effects
6. History of bariatric surgery or currently on weight loss drugs.
7. Uncontrolled hypertension (BP>140/90)
8. Subjects with secondary causes of hypertriglyceridemia: alcoholism, dysglobulinemia, thyroid disease that is poorly controlled (TSH<0.35 or TSH>5.5)
9. Subjects with an abnormal level of liver enzymes (twice the normal level)
10. Suffered from ischemic event such as myocardial infarction, cerebrovascular accident and angina pectoris in the last 6 months
11. Uncontrolled endocrine or metabolic disease known to influence serum lipids or lipoproteins such as cushing syndrome
12. Gastrointestinal disease that may influence lipid metabolism such as celiac, crohn, colitis or other malabsorption problem
13. Subjects who have had any malignancy. Subjects who have had basal cell carcinoma that have been disease free for at least 3 years are eligible for the study.
14. Consumption of one fish serving (200 grams) or sea food x2 a week or more.
15. HIV infection by history
16. History of hypersensitivity or allergy to fish, fish oil or soy
17. BMI≥35
18. Weight change > 3 kg during the run-in period
19. Any other reason that, in the opinion of the investigator, prevents the subject from participating in the study or compromise the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2012-10; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
fasting triglycerides levels | 12 weeks
  Noninferiority of phytosterol esters of omega-3 in affecting plasma fasting triglyceride levels in comparison with Omega-3 acids ethyl esters.

SECONDARY OUTCOMES:
Difference between phytosterol esters of omega-3 and Omega-3 acids ethyl esters treatment groups in other lipid and biomarker levels | 12 weeks
  Difference between phytosterol esters of omega-3 and Omega-3 acids ethyl esters treatment groups in other lipid and biomarker levels

CONTACTS AND LOCATIONS:
Overall Officials: Yossi Azuri, MD, Principal Investigator — Maccabi Healthcare Services, Israel
Locations (1):
- Maccabi Healthcare Services, Tel Aviv, Israel